CLINICAL TRIAL: NCT03340883
Title: A Phase 1/2, Dose Escalation, Safety and Tolerability Study of BION-1301 in Adults With Relapsed or Refractory Multiple Myeloma
Brief Title: Safety and Tolerability of BION-1301 in Adults With Relapsed or Refractory Multiple Myeloma (MM)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No objective responses observed following completion of Phase 1 dose-escalation
Sponsor: Chinook Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADU-CL-16
Record Dates: First submitted 2017-11-03; First posted 2017-11-14 (Actual); Results first posted 2020-09-07 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: Single arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BION-1301 (Experimental): BION-1301 will be administered once every 2 weeks as an intravenous (IV) infusion.
  Interventions: Biological: BION-1301

INTERVENTIONS:
Biological: BION-1301 — a solution for intravenous (IV) administration, diluted and administered Q2W

SUMMARY:
This is a Phase 1/2 study designed to evaluate the safety and tolerability of BION-1301 in adults with relapsed or refractory multiple myeloma whose disease has progressed after 3 or more prior systemic therapies.

DETAILED DESCRIPTION:
An open-label, multi-center, dose-selection Phase 1/2 study (also referred to as ADU-CL-16) evaluating BION-1301, a humanized monoclonal antibody directed against APRIL for the treatment of relapsed or refractory MM. This first-in-human study is designed to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics and initial clinical activity of BION-1301 administered as a single agent.

The study will be conducted in 2 parts. Phase 1 is dose escalation and seeks to determine the recommended phase 2 dose (RP2D). Once an RP2D is identified, Phase 2 of the study will open and continue to evaluate the safety and preliminary efficacy of BION-1301 administered at selected dose level(s).

The population for this study will consist of adults with relapsed or refractory MM whose disease has progressed after at least 3 prior systemic therapies. BION-1301 will be administered in 28-day cycles; the dosing interval will be once every two weeks (Q2W).

ELIGIBILITY:
Key Inclusion Criteria:

Individuals eligible to participate in this study must meet the following key criteria and additional criteria as specified in the protocol:

1. Male or female, aged ≥ 18 years
2. Confirmed diagnosis of MM per IMWG criteria
3. Measurable disease as defined by one or more of the following:

   * Serum M-protein ≥ 0.5 g/dL
   * Urine M-protein ≥ 200 mg/24 hours
   * Serum Free Light Chain (FLC) assay: involved FLC level ≥ 10 mg/dL provided serum FLC ratio is abnormal
   * In cases where SPEP is unreliable, serum quantitative immunoglobulin (qIgA) ≥ 750 mg/dL (0.75 g/dL) is acceptable
4. Relapsed or refractory (Rajkumar, 2011) to 3 or more different prior lines of therapy for MM, including immunomodulatory drugs (IMiDs), proteasome inhibitors (PIs), chemotherapies, or monoclonal antibodies, and not a candidate for, or intolerant to established therapy known to provide clinical benefit.
5. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 - 1
6. Adequate organ and marrow function at Screening, as defined by the study protocol.

Key Exclusion Criteria:

1. Monoclonal gammopathy of undetermined significance (MGUS), smoldering myeloma, Waldenstrom's macroglobulinemia, or IgM myeloma
2. Active plasma cell leukemia (˃ 2.0 × 109/L circulating plasma cells by standard differential)
3. POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)
4. Prior treatment directed to B-cell Activating Factor (BAFF; BLyS), B-cell Maturation Antigen (BCMA;TNFSF17) or Transmembrane Activator and CAML interactor (TACI; TNFSF13B), including antibodies or BCMA- or TACI-directed Chimeric Antigen Receptor (CAR)-T cell therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2019-06-13 (Actual); Study Completion 2019-07-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - James R. Berenson, MD, Inc, West Hollywood, California
  - Winship Cancer Institute/Emory University, Atlanta, Georgia
  - Ohio State University Wexner Medical Center James Cancer Hospital, Columbus, Ohio
  - UPMC (University of Pittsburgh Medical Center) Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Swedish Medical Center, Seattle, Washington
  - Froedtert Hospital & The Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rajkumar SV, Harousseau JL, Durie B, Anderson KC, Dimopoulos M, Kyle R, Blade J, Richardson P, Orlowski R, Siegel D, Jagannath S, Facon T, Avet-Loiseau H, Lonial S, Palumbo A, Zonder J, Ludwig H, Vesole D, Sezer O, Munshi NC, San Miguel J; International Myeloma Workshop Consensus Panel 1. Consensus recommendations for the uniform reporting of clinical trials: report of the International Myeloma Workshop Consensus Panel 1. Blood. 2011 May 5;117(18):4691-5. doi: 10.1182/blood-2010-10-299487. Epub 2011 Feb 3. PMID 21292775

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject enrollment was stopped prematurely due to the sponsor's decision to terminate the study. Therefore, the study did not proceed to the Phase 2 portion of the study protocol. All reporting groups are for Phase 1 only.
Groups:
- BION-1301 50 mg Q2W: 50 mg BION-1301 will be administered once every 2 weeks as an intravenous (IV) infusion.
- BION-1301 150 mg Q2W: 150 mg BION-1301 will be administered once every 2 weeks as an IV infusion.
- BION-1301 450 mg Q2W: 450 mg BION-1301 will be administered once every 2 weeks as an IV infusion.
- BION-1301 1350 mg Q2W: 1350 mg BION-1301 will be administered once every 2 weeks as an IV infusion.
- BION-1301 2700 mg Q2W: 2700 mg BION-1301 will be administered once every 2 weeks as an IV infusion.
- BION-1301 1350 mg QW*8W->Q2W: 1350 mg BION-1301 will be administered as an IV infusion once per week for up to 8 weeks, followed by dosing once every 2 weeks.
Period: Overall Study
Arm/Group | BION-1301 50 mg Q2W | BION-1301 150 mg Q2W | BION-1301 450 mg Q2W | BION-1301 1350 mg Q2W | BION-1301 2700 mg Q2W | BION-1301 1350 mg QW*8W->Q2W
Started | 4 | 3 | 4 | 4 | 3 | 3
Completed | 4 | 3 | 4 | 4 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Phase 1 BION-1301: BION-1301 will be administered once every 2 weeks as an intravenous (IV) infusion.
  BION-1301: a solution for intravenous (IV) administration, diluted and administered Q2W
Arm/Group | Phase 1 BION-1301
Number analyzed (Participants) | 21
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 6
  >=65 years | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 16
  More than one race | 0
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Safety (Phase 1)
Description: Number of patients reporting treatment-related adverse events that qualify as dose-limiting toxicities (DLTs) of BION-1301 as a single agent
Time Frame: 28 days following first administration of BION-1301
Population: Safety Analysis Set (all participants who received any amount of study drug) in the Phase 1 part of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | BION-1301 50 mg Q2W | BION-1301 150 mg Q2W | BION-1301 450 mg Q2W | BION-1301 1350 mg Q2W | BION-1301 2700 mg Q2W | BION-1301 1350 mg QW*8W->Q2W
Number analyzed (Participants) | 4 | 3 | 4 | 4 | 3 | 3
Participants | 0 | 0 | 0 | 1 | 0 | 0

2. Primary Outcome: Recommended Phase 2 Dose (Phase 1)
Description: Recommended Phase 2 Dose RP2D of BION-1301 when administered as a single-agent
Time Frame: Approximately 2 years
Population: Study was terminated early. No outcome measures were assessed.
Arm/Group | BION-1301 50 mg Q2W | BION-1301 150 mg Q2W | BION-1301 450 mg Q2W | BION-1301 1350 mg Q2W | BION-1301 2700 mg Q2W | BION-1301 1350 mg QW*8W->Q2W
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Biomarkers (Phase 1 and 2)
Description: Biomarkers such as soluble a proliferation inducing ligand (APRIL; TNFSF13); soluble B cell maturation antigen (BCMA; TNFRSF17)
Time Frame: Baseline and approximately 2 years
Population: Study was terminated early and Phase 2 did not enroll. BCMA was an exploratory endpoint and was not reported.
Measure: Median (Full Range); unit: % change relative to baseline
Arm/Group | BION-1301 50 mg Q2W | BION-1301 150 mg Q2W | BION-1301 450 mg Q2W | BION-1301 1350 mg Q2W | BION-1301 2700 mg Q2W | BION-1301 1350 mg QW*8W->Q2W
Number analyzed (Participants) | 4 | 3 | 4 | 4 | 3 | 3
% change relative to baseline
  Free APRIL target engagement (AUEC1-15d) | 1000 [580 to 1500] | 970 [750 to 1200] | 470 [190 to 620] | 140 [79 to 510] | 72 [70 to 250] | 200 [56 to 240]
  BCMA: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Bioanalytical Measures (Phase 1 and Phase 2)
Description: Relative change in serum and urine M-protein levels defined as the maximum reduction from baseline
Time Frame: Baseline and approximately 2 years
Population: Some laboratory tests were not performed for some of the participants. Therefore, the number analyzed does not always match the overall number of participants analyzed. Study was terminated early and Phase 2 did not enroll.
Measure: Median (Inter-Quartile Range); unit: percentage change
Arm/Group | BION-1301 50 mg Q2W | BION-1301 150 mg Q2W | BION-1301 450 mg Q2W | BION-1301 1350 mg Q2W | BION-1301 2700 mg Q2W | BION-1301 1350 mg QW*8W->Q2W
Number analyzed (Participants) | 4 | 3 | 4 | 4 | 3 | 3
percentage change
  Serum A/G Ratio (RATIO): number analyzed (Participants) | 2 | 2 | 1 | 0 | 2 | 0
  Serum A/G Ratio (RATIO) | 24.763 [18.182 to 31.343] | 31.538 [23.077 to 40.000] | 28.571 [28.571 to 28.571] |  | 20.202 [18.182 to 22.222] |
  Serum Albumin (g/dL): number analyzed (Participants) | 2 | 3 | 2 | 4 | 3 | 1
  Serum Albumin (g/dL) | 40.191 [27.326 to 53.056] | 5.405 [5.217 to 28.000] | 10.591 [6.897 to 14.286] | 9.294 [3.808 to 17.042] | 3.571 [2.778 to 13.587] | 7.979 [7.979 to 7.979]
  Serum Alpha-1 Globulin (g/dL): number analyzed (Participants) | 2 | 1 | 2 | 1 | 1 | 3
  Serum Alpha-1 Globulin (g/dL) | 18.698 [14.815 to 22.581] | 30.556 [30.556 to 30.556] | 29.710 [26.087 to 33.333] | 24.138 [24.138 to 24.138] | 16.129 [16.129 to 16.129] | 20.000 [18.919 to 50.000]
  Serum Alpha-2 Globulin (g/dL): number analyzed (Participants) | 3 | 1 | 3 | 3 | 1 | 3
  Serum Alpha-2 Globulin (g/dL) | 2.985 [2.439 to 20.408] | 31.579 [31.579 to 31.579] | 14.286 [13.415 to 14.754] | 10.843 [9.756 to 12.037] | 14.286 [14.286 to 14.286] | 10.000 [4.918 to 33.333]
  Serum Beta Globulin (g/dL): number analyzed (Participants) | 1 | 1 | 1 | 1 | 2 | 1
  Serum Beta Globulin (g/dL) | 33.636 [33.636 to 33.636] | 3.125 [3.125 to 3.125] | 0.542 [0.542 to 0.542] | 22.472 [22.472 to 22.472] | 8.571 [7.143 to 10.000] | 2.609 [2.609 to 2.609]
  Serum Gamma Globulin (g/dL): number analyzed (Participants) | 3 | 1 | 3 | 2 | 1 | 0
  Serum Gamma Globulin (g/dL) | 13.920 [8.511 to 41.667] | 96.552 [96.552 to 96.552] | 25.926 [15.789 to 50.000] | 23.441 [22.807 to 24.074] | 0.627 [0.627 to 0.627] |
  Serum Immunoglobulin A (g/L): number analyzed (Participants) | 1 | 1 | 2 | 2 | 3 | 1
  Serum Immunoglobulin A (g/L) | 1.615 [1.615 to 1.615] | 66.667 [66.667 to 66.667] | 36.174 [0.717 to 71.631] | 30.536 [12.500 to 48.571] | 23.077 [16.667 to 70.588] | 23.077 [23.077 to 23.077]
  Serum Immunoglobulin G (g/L): number analyzed (Participants) | 2 | 2 | 2 | 2 | 0 | 1
  Serum Immunoglobulin G (g/L) | 25.274 [8.312 to 42.236] | 25.000 [16.788 to 33.212] | 25.016 [22.566 to 27.467] | 20.125 [14.888 to 25.362] |  | 0.352 [0.352 to 0.352]
  Serum Immunoglobulin M (g/L): number analyzed (Participants) | 3 | 3 | 1 | 2 | 2 | 0
  Serum Immunoglobulin M (g/L) | 27.273 [27.273 to 76.563] | 28.571 [14.286 to 40.000] | 40.000 [40.000 to 40.000] | 61.364 [54.545 to 68.182] | 64.148 [46.154 to 82.143] |
  Serum Kappa Light Chain, Free (mg/dL): number analyzed (Participants) | 3 | 1 | 2 | 2 | 1 | 2
  Serum Kappa Light Chain, Free (mg/dL) | 34.0000 [6.7568 to 46.4419] | 5.9735 [5.9735 to 5.9735] | 42.0349 [30.0000 to 54.0698] | 72.4863 [69.3627 to 75.6098] | 64.8649 [64.8649 to 64.8649] | 47.9787 [30.0000 to 65.9574]
  Serum Kappa LtChain,Free/LambdaLtChain,Free(RATIO): number analyzed (Participants) | 2 | 0 | 1 | 2 | 1 | 1
  Serum Kappa LtChain,Free/LambdaLtChain,Free(RATIO) | 53.919 [50.000 to 57.838] |  | 50.000 [50.000 to 50.000] | 100.000 [100.000 to 100.000] | 60.000 [60.000 to 60.000] | 100.000 [100.000 to 100.000]
  Serum Lambda Light Chain, Free (mg/dL): number analyzed (Participants) | 2 | 2 | 3 | 2 | 2 | 0
  Serum Lambda Light Chain, Free (mg/dL) | 13.9651 [7.0000 to 20.9302] | 26.3520 [11.1111 to 41.5929] | 13.4372 [13.4028 to 57.6642] | 26.9335 [12.5000 to 41.3669] | 24.5619 [20.0000 to 29.1237] |
  Serum Monoclonal Protein Spike (g/dL): number analyzed (Participants) | 3 | 0 | 1 | 1 | 0 | 0
  Serum Monoclonal Protein Spike (g/dL) | 13.1579 [1.0526 to 50.0000] |  | 5.4670 [5.4670 to 5.4670] | 27.2727 [27.2727 to 27.2727] |  |
  Serum Protein (g/dL): number analyzed (Participants) | 1 | 0 | 2 | 1 | 1 | 2
  Serum Protein (g/dL) | 8.14 [8.14 to 8.14] |  | 3.06 [2.88 to 3.23] | 3.03 [3.03 to 3.03] | 6.74 [6.74 to 6.74] | 3.05 [1.69 to 4.41]
  Urine Albumin (mg/dL): number analyzed (Participants) | 0 | 1 | 0 | 0 | 2 | 0
  Urine Albumin (mg/dL) |  | 18.1818 [18.1818 to 18.1818] |  |  | 54.7349 [20.6055 to 88.8643] |
  Urine Alpha-1 Globulin (mg/dL): number analyzed (Participants) | 0 | 1 | 0 | 0 | 2 | 0
  Urine Alpha-1 Globulin (mg/dL) |  | 80.0000 [80.0000 to 80.0000] |  |  | 71.7418 [60.4982 to 82.9854] |
  Urine Alpha-2 Globulin (mg/dL): number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 0
  Urine Alpha-2 Globulin (mg/dL) |  |  |  |  | 63.5621 [37.2727 to 89.8515] |
  Urine Beta Globulin (mg/dL): number analyzed (Participants) | 0 | 0 | 0 | 1 | 2 | 0
  Urine Beta Globulin (mg/dL) |  |  |  | 19.4996 [19.4996 to 19.4996] | 49.3411 [6.6748 to 92.0074] |
  Urine Gamma Globulin (mg/dL): number analyzed (Participants) | 0 | 1 | 1 | 0 | 1 | 0
  Urine Gamma Globulin (mg/dL) |  | 90.3185 [90.3185 to 90.3185] | 100.0000 [100.0000 to 100.0000] |  | 93.1735 [93.1735 to 93.1735] |
  Urine Monoclonal Protein Spike (%): number analyzed (Participants) | 0 | 0 | 0 | 1 | 1 | 1
  Urine Monoclonal Protein Spike (%) |  |  |  | 2.755 [2.755 to 2.755] | 30.695 [30.695 to 30.695] | 11.819 [11.819 to 11.819]
  Urine Protein (mg/dL): number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 0
  Urine Protein (mg/dL) |  |  |  |  | 52.9665 [14.2857 to 91.6472] |
  Urine Protein, Calculated (mg/24hr): number analyzed (Participants) | 0 | 0 | 1 | 0 | 2 | 0
  Urine Protein, Calculated (mg/24hr) |  |  | 9.1743 [9.1743 to 9.1743] |  | 42.9298 [15.0943 to 70.7652] |

5. Primary Outcome: Safety Profile (Phase 2)
Description: BION-1301 safety profile based on incidence of TEAEs (treatment emergent adverse events), changes in safety parameters, and unacceptable toxicities
Time Frame: 28 days
Population: Study was terminated early and Phase 2 was not enrolled. Safety profile was not assessed.
Arm/Group | BION-1301 50 mg Q2W | BION-1301 150 mg Q2W | BION-1301 450 mg Q2W | BION-1301 1350 mg Q2W | BION-1301 2700 mg Q2W | BION-1301 1350 mg QW*8W->Q2W
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Response Rate (Phase 2)
Description: Objective response rate (ORR) based on International Myeloma Working Group (IMWG) uniform response criteria of stringent complete response (sCR), complete response (CR), very good partial response (VGPR), or partial response (PR)
Time Frame: Approximately 30 months
Population: Study was terminated early and Phase 2 was not enrolled. Objective response rate was not assessed.
Arm/Group | BION-1301 50 mg Q2W | BION-1301 150 mg Q2W | BION-1301 450 mg Q2W | BION-1301 1350 mg Q2W | BION-1301 2700 mg Q2W | BION-1301 1350 mg QW*8W->Q2W
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Progression-Free Survival (Phase 2)
Description: Progression-free survival (PFS) defined as time from first dose of study drug to date of first tumor progression or death due to any cause
Time Frame: Approximately 30 months
Population: Study was terminated early and Phase 2 did not enroll. Progression-free survival was not assessed.
Arm/Group | BION-1301 50 mg Q2W | BION-1301 150 mg Q2W | BION-1301 450 mg Q2W | BION-1301 1350 mg Q2W | BION-1301 2700 mg Q2W | BION-1301 1350 mg QW*8W->Q2W
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Overall Survival (Phase 2)
Description: Overall survival (OS) defined as the time from first dose of study drug to date of death due to any cause
Time Frame: Approximately 30 months
Population: Study was terminated early and Phase 2 did not enroll. Overall survival was not assessed.
Arm/Group | BION-1301 50 mg Q2W | BION-1301 150 mg Q2W | BION-1301 450 mg Q2W | BION-1301 1350 mg Q2W | BION-1301 2700 mg Q2W | BION-1301 1350 mg QW*8W->Q2W
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the start of the first study drug administration until 28 days after the last study drug dose, assessed up to 1 year from the date of randomization.
Arm/Group | BION-1301 50 mg Q2W | BION-1301 150 mg Q2W | BION-1301 450 mg Q2W | BION-1301 1350 mg Q2W | BION-1301 2700 mg Q2W | BION-1301 1350 mg QW*8W->Q2W
All-Cause Mortality (participants affected / at risk) | 1/4 | 2/3 | 0/4 | 2/4 | 1/3 | 1/3
Serious Adverse Events (participants affected / at risk) | 3/4 | 1/3 | 1/4 | 2/4 | 0/3 | 1/3
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 4/4 | 3/4 | 2/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BION-1301 50 mg Q2W (N=4) | BION-1301 150 mg Q2W (N=3) | BION-1301 450 mg Q2W (N=4) | BION-1301 1350 mg Q2W (N=4) | BION-1301 2700 mg Q2W (N=3) | BION-1301 1350 mg QW*8W->Q2W (N=3)
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Sudden death (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BION-1301 50 mg Q2W (N=4) | BION-1301 150 mg Q2W (N=3) | BION-1301 450 mg Q2W (N=4) | BION-1301 1350 mg Q2W (N=4) | BION-1301 2700 mg Q2W (N=3) | BION-1301 1350 mg QW*8W->Q2W (N=3)
Constipation (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 3 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 0 | 1 | 1 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Localised oedema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Rhinovirus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 2 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 2 | 1 | 1
Hypotension (Vascular disorders) | 1 | 0 | 0 | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Muscle spasticity (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood fibrinogen decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Head and neck cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
ADU-CL-16 was terminated early leading to a small number of Phase 1 subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosure restriction - study results first published in a joint multi-center paper unless (a) no multi-center publication, or (b) ≥18 months has passed since completion of the study. Thereafter, Investigator may publish provided that Investigator: (i) provides a copy of the publication to Aduro ≥ 60 days in advance of submission for publication; (ii) deletes Aduro Confidential Information (other than the Study results) and (iii) submission may be delayed up to 90 days to permit IP filings.

DOCUMENTS (2):
  • Study Protocol (2018-11-13): https://cdn.clinicaltrials.gov/large-docs/83/NCT03340883/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-18): https://cdn.clinicaltrials.gov/large-docs/83/NCT03340883/SAP_001.pdf